CLINICAL TRIAL: NCT04764201
Title: A Randomized, Open Label, Single Dose, 2-way Crossover Clinical Trial to Evaluate the Pharmacokinetic Characteristics and Safety Between HIP2001 and HGP2001 in Healthy Volunteers
Brief Title: The Pharmacokinetic Characteristics and Safety Between HIP2001 and HGP2001 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HM-EDOX-101
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Other): Period 1: HGP2001, Period 2: HIP2001
  Interventions: Drug: HIP2001; Drug: HGP2001
- Sequence 2 (Other): Period 1: HIP2001, Period 2: HGP2001
  Interventions: Drug: HIP2001; Drug: HGP2001

INTERVENTIONS:
Drug: HIP2001 — Test drug
Drug: HGP2001 — Reference drug

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetic characteristics and safety between HIP2001 and HGP2001 in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* 19 kg/m^2 ≤ BMI < 28 kg/m^2, weight >60kg
* 90 mmHg ≤ SBP <140 mmHg, 50 mmHg ≤ DBP <900 mmHg
* agrees that the person, spouse, or partner uses appropriate medically recognized contraception and does not provide sperm or eggs from the date of administration of the first investigational drug to 7 days after the administration of the last investigational drug.

Exclusion Criteria:

* A history of hypersensitivity reactions or clinically significant hypersensitivity reactions
* A history of gastrointestinal diseases or surgery that may affect the absorption of clinical trial drugs
* A history of substance abuse or who test positive for drugs of concern for abuse in the urine drug screening test
* Positive results of serological tests
* Have taken other investigational drugs or bioequivalence drugs within 6 months before the first administration of the investigational drug
* Donated whole blood within 60 days prior to the screening date or donated components within 30 days or received a blood transfusion within 30 days
* Have drank more than 210 g/week of alcohol within 30 days before the screening date
* Have smoked more than 10 bills/day within 30 days before the screening date
* AST, ALT value is more than 2 times the UNL or bilirubin level is more than 1.5 times the UNL, eGFR < 50 mL/min/1.73m2, Prothrombin (INR) > 1.31 INR or aPTT > 39.7 sec
* 12-ECG QTc >450 ms

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2021-01-16 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-03-08 (Actual)

PRIMARY OUTCOMES:
AUCt | 0~48 hours
  Pharmacokinetic evaluation
Cmax | 0~48 hours
  Pharmacokinetic evaluation

SECONDARY OUTCOMES:
AUCinf | 0~48 hours
  Pharmacokinetic evaluation
Tmax | 0~48 hours
  Pharmacokinetic evaluation
t1/2 | 0~48 hours
  Pharmacokinetic evaluation
CL/F | 0~48 hours
  Pharmacokinetic evaluation
Vd/F | 0~48 hours
  Pharmacokinetic evaluation

CONTACTS AND LOCATIONS:
Overall Officials: Mingeul Kim, Principal Investigator — Jeonbuk University Hospital
Locations (1):
- Jeonbuk University Hospital, Jeonju, South Korea